CLINICAL TRIAL: NCT04971278
Title: Evaluating the Impact of a Supportive Care Program
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: QI-High Risk
Record Dates: First submitted 2021-07-14; First posted 2021-07-21 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Patient Engagement; Morality
MeSH Terms: conditions — Patient Participation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- HealthFirst Intervention: Patients attributed to HealthFirst who will receive the intervention
  Interventions: Behavioral: Supportive care program
- HealthFirst Control: Patients attributed to HealthFirst who will not receive the intervention
- Mortality Model Intervention: Patients who are identified as High Risk by the mortality predictive model and who receive the intervention.
  Interventions: Behavioral: Supportive care program
- Mortality Model Control: Patients who are identified as High Risk by the mortality predictive model and who do not receive the intervention.

INTERVENTIONS:
Behavioral: Supportive care program — Community Health Workers, a home visiting doctor service, a supportive care nurse, and behavioral health specialist engage the population to address a range of biopsychosocial needs with end goal in increasing support in the community and engaging palliative and hospice care when appropriate to prevent hospital readmissions, shorten length of stay, reduce hospital utilization, and decrease overall patient cost with a focus on hospital spend.
  Groups: HealthFirst Intervention; Mortality Model Intervention

SUMMARY:
NYU's High Risk Program targets patients who may be more likely to have increased hospitalization due to health conditions that may cause death in the near future. Community Health Workers, a home visiting doctor service, a supportive care nurse, and behavioral health specialist engage the population to address a range of biopsychosocial needs with end goal in increasing support in the community and engaging palliative and hospice care when appropriate to prevent hospital readmissions, shorten length of stay, reduce hospital utilization, and decrease overall patient cost with a focus on hospital spend.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* at or above the 75th percentile on the Mortality Model
* Attributed to a value based contract

Exclusion Criteria:

* Less than 18 years of age
* Below the 75th percentile on the Mortality Model
* Not attributed to a value based contract

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: NYU Langone adult patients (>18 years old) at or above the 75th percentile on NYU's mortality model currently attributed to one of DSRIP's value based contracts.
Sampling Method: Probability Sample
Enrollment: 1201 (Actual)
Dates: Start 2019-11-07 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-09-22 (Actual)

PRIMARY OUTCOMES:
Rate of Advance Care Planning note creation | 2 years
  How many and how often are ACP notes written for patients

CONTACTS AND LOCATIONS:
Overall Officials: Leora Horwitz, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States